CLINICAL TRIAL: NCT03392324
Title: Feasibility Study of Compensation for Blindness With the PRIMA System in Patients With Atrophic Dry Age Related Macular Degeneration
Brief Title: PRIMA US-Feasibility Study in Atrophic Dry AMD
Acronym: PRIMA-FS-US
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-PRIMA-FS-US
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: atrophic macular degeneration; geographic atrophy; retina implant; retinal prosthesis; visual prosthesis; macular degeneration; dry macular degeneration; AMD
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PRIMA (Experimental): Implantation of PRIMA device
  Interventions: Device: PRIMA

INTERVENTIONS:
Device: PRIMA — Implantation of PRIMA device

SUMMARY:
In this early feasibility trial the safety and performance of the new retinal prothesis PRIMA is tested in five subjects suffering from atrophic dry age related macular degeneration.

DETAILED DESCRIPTION:
PRIMA is a new photovoltaic sub-retinal wireless prosthesis for partial restoration of visual perception in patients with vision loss from atrophic dry Age-related Macular Degeneration. The implantable part of the device is placed under the retina. A mini camera mounted on a pair of glasses captures the visual scene in the environment. The visual scene is processed and simplified by the pocket computer connected to the glasses in order to extract useful information from the images. The simplified images are then sent back to the glasses where a miniaturized projector then projects the processed images wirelessly via pulses of near infrared light on the PRIMA implant at the back of the eye under the retina. The photovoltaic cells convert this optical information into electrical stimulation to excite the nerve cells of the retina and induce visual perception. In this early feasibility study five human subjects suffering from atrophic dry age related macular degeneration will receive the implant. The performance and the safety of the device will be monitored for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Is 60 years or older at the date of inclusion;
* Has a confirmed diagnosis of atrophic dry age related macular degeneration with an atrophy size of at least 3 optic disc diameters in the study eye;
* Has best corrected visual acuity of logMAR 1.3 (20/400) or worse in the study eye measured by ETDRS;
* Has a central scotoma in the study eye with no perception at 0 dB on MP-1 micro-perimetry scale in the visual field covering the central 7 degrees (+/-3.5 degrees) and maximum 20% perception in the remaining visual field covering the central 12 degrees (+/- 6 degrees);
* Meets one of the following criteria in the non-study eye:

  * Visual acuity of 20/200 (logMAR 1.0) or worse and an atrophy size <8mm2
  * Visual acuity of 20/160 (logMAR 0.9) or worse and an atrophy size ≥8mm2 and ≤12.5 mm2
  * Visual acuity of 20/100 (logMAR 0.7) or worse and an atrophy size >12.5 mm2
* Has a refraction of study eye between -3 and + 4 (limits included) for patients with IOL (there is no refraction criteria for phakic patients);
* Understands and accepts the obligation to present for all schedule follow-up visits;
* Patient signed informed consent.

Main Exclusion Criteria:

* Has cataract in the study ;
* Has an aphakic study eye;
* Has no light perception in the study eye;
* Has a history of choroidal neovascularization in either eye;
* Has any disease (other than study allowed diseases) or condition that affects retinal function of the study eye
* Has an implanted telescope in one eye;
* Has any disease or condition that prevents adequate examination of the study
* Has a corneal endothelial cell count of less than 1000 cells/mm² in the study eye
* Suffers from nystagmus or other ocular motility disorders;
* Has any disease or condition that precludes the understanding or communication of the informed consent, study requirements or test protocols
* Has a history of epileptic seizure;
* Has a history of chronic or recurrent infection or inflammation that would preclude participation in the study;
* Presents with hypotony or hypertony in the study eye;
* Has another active implanted device;
* Has active cancer or a history of intraocular, optic nerve or brain cancer and metastasis;
* Is an immune-suppressed subject;
* Is carrier of multi-resistant microorganisms;
* Is receiving anticoagulation therapy that cannot be adapted to allow eye surgery;
* Is participating in another investigational drug or device study that may interfere with the present study;
* Has recurrent or chronic inflammations or infections;
* Has a severe psychological disorder;
* Does not have the mental capacity to legally sign the informed consent;
* Has severe renal, cardiac, hepatic, etc. organ diseases;
* Has head dimensions that are incompatible with the Visual Interface;
* Has too high and unrealistic expectation;

Detailed patient criteria will be verified by the study doctor.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Near Visual Acuity | 12 months after implantation
  Near Visual acuity measured by FrACT

SECONDARY OUTCOMES:
Near Visual Acuity | 3, 6, 9, 18, 24, and 36 months after implantation
  Near Visual acuity measured by FrACT
Visual Acuity | 3, 6, 9, 12, 18, 24 and 36 months after implantation
  Visual acuity measured by ETDRS
Reading Acuity Test | 6, 12, 24, 36 months after implantation
  Reading acuity measured by Radner Charts
Quality of Life | 12, 24, and 36 months after implantation
  The change in quality of life is measure by the Impact of Vision Impairment (IVI) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Martel, MD, Principal Investigator — UPMC Pittsburgh
Locations (3):
- United States (3):
  - Byers Eye Institute-Stanford University, Palo Alto, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - UPMC Eye Center, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Pixium Vision — http://www.pixium-vision.com